CLINICAL TRIAL: NCT02360696
Title: Predictors of Clinical Response to Montelukast in Children With Functional Dyspepsia
Brief Title: Functional Dyspepsia (FD) - Clinical Response to Montelukast in Children
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Craig A. Friesen, MD, Section Chief/Division of Gastroenteroly, Hepatology, and Nutrition, Children's Mercy Hospital Kansas City
Other Study IDs: 13100348
Record Dates: First submitted 2014-09-03; First posted 2015-02-11 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Eosinophilia; Dyspepsia
Keywords: Duodenal Eosinophilia; Functional Dyspepsia; Mucosal Eosinophilia
MeSH Terms: conditions — Eosinophilia; Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained, with potential for extraction of DNA from at least one of the types of samples retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peds/Adol Pts w/ FD - CMH GI APT clinic: Phase 1. Standard-of-Care Endoscopy to establish baseline data and immunohistochemistry studies. Additional biopsies taken for DNA and microarray analysis. If participant biopsies meet criteria (> or = 20/hpf) and no nodularity or tumors, s/he will be eligible to move to second phase.
  Phase 2. Standard of care treatment of 3 mg/kg ranitidine bid and 20 mg. montelukast each AM for three weeks. Based on response to global assessment score, participants will be placed in non-responder or responder group. Participants from the responder group will move to final phase of the study.
  Phase 3: Research endoscopy to measure response to montelukast therapy. Biopsies taken for cell density counts and immunohistochemistry studies. Additional biopsies taken for DNA and microarray analysis.

SUMMARY:
Duodenal eosinophilia has been associated with dyspepsia in adults and the investigators have previously described the finding of duodenal mucosal eosinophilia in 71-79% of children undergoing diagnostic endoscopy. Previous studies in children have shown positive response to montelukast with approximately 50% finding complete relief and 20-30 percent showing no response.

There are a number of factors that have the potential to contribute to the observed variability in response to montelukast. These include variability in:

1. systemic drug exposure (drug absorption, biotransformation and/or elimination)
2. regulation of leukotriene biosynthesis
3. cysteinyl leukotriene receptors and downstream mediators
4. patient disease phenotype (e.g. Functional Gastrointestinal Disorder (FGID) disease classification, psychologic profile)

In this study, the investigators propose to utilize biopsy specimens stratified by drug response to identify candidate gene expression modules that will be validated in a prospective study design. The overall goal of this program is to develop a signature of montelukast response that can be applied not only to eosinophilic gastroenteritis, but more generally to other diseases, such as asthma, where the drug is widely used with variable success.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 - 17 years, inclusive
* Abdominal pain of at least 8 weeks duration and fulfilling symptom- based criteria for functional dyspepsia
* Scheduled for endoscopy following failure to respond to acid-reduction therapy
* Evidence of written parental permission (consent) and subject assent

Exclusion Criteria:

* Previous treatment with montelukast
* Treatment with corticosteroids or oral cromolyn sodium in the four weeks prior to enrollment
* Prior history or clinical signs/symptoms of chronic disease requiring regular medical care (e.g., diabetes mellitus, juvenile idiopathic arthritis, cystic fibrosis or cancer)
* Exposure within the past two weeks to drugs or natural products that induce CYP2C8/9 or CYP3A4, including amprenavir, carbamazepine, lopinavir/ritonavir, nafcillin, nevirapine, oxcarbazepine, phenobarbital, phenytoin, rifampin, St. John's Wort, or that inhibit CYP2C8/9 or CYP3A4, such as ciprofloxacin, clarithromycin, erythromycin, fluconazole, fluvoxamine, grapefruit juice, paroxetine, sertraline, sulfamethoxazole, trimethoprim
* A Body Mass Index of 30 or greater
* Non-English speaking
* Those patients who will turn 18 during the duration of the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Up to 50 subjects (allowance of 20 additional subjects for screen fails and those who will not complete Phase 3 of the study) will be recruited from a cohort of patients referred to the Abdominal Pain Clinic at Children's Mercy Hospitals and Clinics and enrolled prior to routine initial endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Identification of a signature of montelukast response using gene expression patterns in biopsy samples from clinical responders and non-responders to montelukast. | Approximately 7-8 weeks
  Identification of patients who will benefit from montelukast therapy , allowing more efficient, and possibly more effective, care.

SECONDARY OUTCOMES:
Characterization a signature of montelukast response using comparison gene expression patterns in biopsy samples obtained before and after montelukast therapy in children with a positive clinical response to the drug. | 7-8 weeks.
  Identification and development of a signature of montelukast response applied to eosinophilic gastroenteritis, and more generally to other diseases, such as asthma, where the drug is widely used with variable success.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Friesen, MD, Principal Investigator — Children's Mercy, Division of Gastroenterlogy, Hepatology, and Nutrition; Steven Leeder, PharmD, PhD, Principal Investigator — Children's Mercy, Division of Clinical Pharmacology and Medical Toxicology
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

REFERENCES:
- [Background] Talley NJ, Walker MM, Aro P, Ronkainen J, Storskrubb T, Hindley LA, Harmsen WS, Zinsmeister AR, Agreus L. Non-ulcer dyspepsia and duodenal eosinophilia: an adult endoscopic population-based case-control study. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1175-83. doi: 10.1016/j.cgh.2007.05.015. Epub 2007 Aug 7. PMID 17686660
- [Background] Friesen CA, Neilan NA, Schurman JV, Taylor DL, Kearns GL, Abdel-Rahman SM. Montelukast in the treatment of duodenal eosinophilia in children with dyspepsia: effect on eosinophil density and activation in relation to pharmacokinetics. BMC Gastroenterol. 2009 May 11;9:32. doi: 10.1186/1471-230X-9-32. PMID 19432972
- [Background] Friesen CA, Sandridge L, Andre L, Roberts CC, Abdel-Rahman SM. Mucosal eosinophilia and response to H1/H2 antagonist and cromolyn therapy in pediatric dyspepsia. Clin Pediatr (Phila). 2006 Mar;45(2):143-7. doi: 10.1177/000992280604500205. PMID 16528434
- [Background] Erjefalt JS, Greiff L, Andersson M, Adelroth E, Jeffery PK, Persson CG. Degranulation patterns of eosinophil granulocytes as determinants of eosinophil driven disease. Thorax. 2001 May;56(5):341-4. doi: 10.1136/thorax.56.5.341. PMID 11312400
- [Background] Friesen CA, Andre L, Garola R, Hodge C, Roberts C. Activated duodenal mucosal eosinophils in children with dyspepsia: a pilot transmission electron microscopic study. J Pediatr Gastroenterol Nutr. 2002 Sep;35(3):329-33. doi: 10.1097/00005176-200209000-00017. PMID 12352522
- [Background] Hall W, Buckley M, Crotty P, O'Morain CA. Gastric mucosal mast cells are increased in Helicobacter pylori-negative functional dyspepsia. Clin Gastroenterol Hepatol. 2003 Sep;1(5):363-9. doi: 10.1053/s1542-3565(03)00184-8. PMID 15017654
- [Background] Friesen CA, Lin Z, Singh M, Singh V, Schurman JV, Burchell N, Cocjin JT, McCallum RW. Antral inflammatory cells, gastric emptying, and electrogastrography in pediatric functional dyspepsia. Dig Dis Sci. 2008 Oct;53(10):2634-40. doi: 10.1007/s10620-008-0207-0. Epub 2008 Mar 5. PMID 18320315
- [Background] Muijsers RB, Noble S. Montelukast: a review of its therapeutic potential in asthma in children 2 to 14 years of age. Paediatr Drugs. 2002;4(2):123-39. doi: 10.2165/00128072-200204020-00005. PMID 11888359
- [Background] Neustrom MR, Friesen C. Treatment of eosinophilic gastroenteritis with montelukast. J Allergy Clin Immunol. 1999 Aug;104(2 Pt 1):506. doi: 10.1016/s0091-6749(99)70404-5. No abstract available. PMID 10452782
- [Background] Schwartz DA, Pardi DS, Murray JA. Use of montelukast as steroid-sparing agent for recurrent eosinophilic gastroenteritis. Dig Dis Sci. 2001 Aug;46(8):1787-90. doi: 10.1023/a:1010682310928. PMID 11508684
- [Background] Vanderhoof JA, Young RJ, Hanner TL, Kettlehut B. Montelukast: use in pediatric patients with eosinophilic gastrointestinal disease. J Pediatr Gastroenterol Nutr. 2003 Feb;36(2):293-4. doi: 10.1097/00005176-200302000-00027. No abstract available. PMID 12548071
- [Background] Friesen CA, Kearns GL, Andre L, Neustrom M, Roberts CC, Abdel-Rahman SM. Clinical efficacy and pharmacokinetics of montelukast in dyspeptic children with duodenal eosinophilia. J Pediatr Gastroenterol Nutr. 2004 Mar;38(3):343-51. doi: 10.1097/00005176-200403000-00021. PMID 15076638
- [Background] Chiba M, Xu X, Nishime JA, Balani SK, Lin JH. Hepatic microsomal metabolism of montelukast, a potent leukotriene D4 receptor antagonist, in humans. Drug Metab Dispos. 1997 Sep;25(9):1022-31. PMID 9311616
- [Background] Karonen T, Filppula A, Laitila J, Niemi M, Neuvonen PJ, Backman JT. Gemfibrozil markedly increases the plasma concentrations of montelukast: a previously unrecognized role for CYP2C8 in the metabolism of montelukast. Clin Pharmacol Ther. 2010 Aug;88(2):223-30. doi: 10.1038/clpt.2010.73. Epub 2010 Jun 30. PMID 20592724
- [Background] Filppula AM, Laitila J, Neuvonen PJ, Backman JT. Reevaluation of the microsomal metabolism of montelukast: major contribution by CYP2C8 at clinically relevant concentrations. Drug Metab Dispos. 2011 May;39(5):904-11. doi: 10.1124/dmd.110.037689. Epub 2011 Feb 2. PMID 21289076
- [Background] Daily EB, Aquilante CL. Cytochrome P450 2C8 pharmacogenetics: a review of clinical studies. Pharmacogenomics. 2009 Sep;10(9):1489-510. doi: 10.2217/pgs.09.82. PMID 19761371
- [Background] Rodriguez-Antona C, Niemi M, Backman JT, Kajosaari LI, Neuvonen PJ, Robledo M, Ingelman-Sundberg M. Characterization of novel CYP2C8 haplotypes and their contribution to paclitaxel and repaglinide metabolism. Pharmacogenomics J. 2008 Aug;8(4):268-77. doi: 10.1038/sj.tpj.6500482. Epub 2007 Oct 9. PMID 17923851
- [Background] Zanger UM, Turpeinen M, Klein K, Schwab M. Functional pharmacogenetics/genomics of human cytochromes P450 involved in drug biotransformation. Anal Bioanal Chem. 2008 Nov;392(6):1093-108. doi: 10.1007/s00216-008-2291-6. Epub 2008 Aug 10. PMID 18695978
- [Background] Mougey EB, Feng H, Castro M, Irvin CG, Lima JJ. Absorption of montelukast is transporter mediated: a common variant of OATP2B1 is associated with reduced plasma concentrations and poor response. Pharmacogenet Genomics. 2009 Feb;19(2):129-38. doi: 10.1097/FPC.0b013e32831bd98c. PMID 19151602
- [Background] Mougey EB, Lang JE, Wen X, Lima JJ. Effect of citrus juice and SLCO2B1 genotype on the pharmacokinetics of montelukast. J Clin Pharmacol. 2011 May;51(5):751-60. doi: 10.1177/0091270010374472. Epub 2010 Oct 25. PMID 20974993
- [Background] Kearns GL, Abdel-Rahman SM, Alander SW, Blowey DL, Leeder JS, Kauffman RE. Developmental pharmacology--drug disposition, action, and therapy in infants and children. N Engl J Med. 2003 Sep 18;349(12):1157-67. doi: 10.1056/NEJMra035092. No abstract available. PMID 13679531
- [Background] Knorr B, Larson P, Nguyen HH, Holland S, Reiss TF, Chervinsky P, Blake K, van Nispen CH, Noonan G, Freeman A, Haesen R, Michiels N, Rogers JD, Amin RD, Zhao J, Xu X, Seidenberg BC, Gertz BJ, Spielberg S. Montelukast dose selection in 6- to 14-year-olds: comparison of single-dose pharmacokinetics in children and adults. J Clin Pharmacol. 1999 Aug;39(8):786-93. doi: 10.1177/00912709922008434. PMID 10434229
- [Background] Duroudier NP, Tulah AS, Sayers I. Leukotriene pathway genetics and pharmacogenetics in allergy. Allergy. 2009 Jun;64(6):823-39. doi: 10.1111/j.1398-9995.2009.02015.x. Epub 2009 Mar 26. PMID 19416143
- [Background] Lima JJ, Zhang S, Grant A, Shao L, Tantisira KG, Allayee H, Wang J, Sylvester J, Holbrook J, Wise R, Weiss ST, Barnes K. Influence of leukotriene pathway polymorphisms on response to montelukast in asthma. Am J Respir Crit Care Med. 2006 Feb 15;173(4):379-85. doi: 10.1164/rccm.200509-1412OC. Epub 2005 Nov 17. PMID 16293801
- [Background] Singh RK, Gupta S, Dastidar S, Ray A. Cysteinyl leukotrienes and their receptors: molecular and functional characteristics. Pharmacology. 2010;85(6):336-49. doi: 10.1159/000312669. Epub 2010 Jun 2. PMID 20516735
- [Background] Lima JJ. Treatment heterogeneity in asthma: genetics of response to leukotriene modifiers. Mol Diagn Ther. 2007;11(2):97-104. doi: 10.1007/BF03256228. PMID 17397245
- [Background] Sampson AP, Pizzichini E, Bisgaard H. Effects of cysteinyl leukotrienes and leukotriene receptor antagonists on markers of inflammation. J Allergy Clin Immunol. 2003 Jan;111(1 Suppl):S49-59; discussion S59-61. doi: 10.1067/mai.2003.24. PMID 12532086
- [Background] Bizzintino JA, Khoo SK, Zhang G, Martin AC, Rueter K, Geelhoed GC, Goldblatt J, Laing IA, Le Souef PN, Hayden CM. Leukotriene pathway polymorphisms are associated with altered cysteinyl leukotriene production in children with acute asthma. Prostaglandins Leukot Essent Fatty Acids. 2009 Jul;81(1):9-15. doi: 10.1016/j.plefa.2009.05.022. Epub 2009 Jun 12. PMID 19524426
- [Background] Bischoff SC, Lorentz A, Schwengberg S, Weier G, Raab R, Manns MP. Mast cells are an important cellular source of tumour necrosis factor alpha in human intestinal tissue. Gut. 1999 May;44(5):643-52. doi: 10.1136/gut.44.5.643. PMID 10205200
- [Background] Peters-Golden M, Gleason MM, Togias A. Cysteinyl leukotrienes: multi-functional mediators in allergic rhinitis. Clin Exp Allergy. 2006 Jun;36(6):689-703. doi: 10.1111/j.1365-2222.2006.02498.x. PMID 16776669
- [Background] Aguillon JC, Cruzat A, Aravena O, Salazar L, Llanos C, Cuchacovich M. Could single-nucleotide polymorphisms (SNPs) affecting the tumour necrosis factor promoter be considered as part of rheumatoid arthritis evolution? Immunobiology. 2006;211(1-2):75-84. doi: 10.1016/j.imbio.2005.09.005. Epub 2005 Dec 27. PMID 16446172
- [Background] de Vries N, Tak PP. The response to anti-TNF-alpha treatment: gene regulation at the bedside. Rheumatology (Oxford). 2005 Jun;44(6):705-7. doi: 10.1093/rheumatology/keh662. Epub 2005 Apr 26. No abstract available. PMID 15855186
- [Background] Maeba S, Ichiyama T, Ueno Y, Makata H, Matsubara T, Furukawa S. Effect of montelukast on nuclear factor kappaB activation and proinflammatory molecules. Ann Allergy Asthma Immunol. 2005 Jun;94(6):670-4. doi: 10.1016/S1081-1206(10)61326-9. PMID 15984600
- [Background] Kim SH, Yang EM, Kim SH, Park HS. Regulation of monocyte chemoattractant protein 1 by cysteinyl leukotriene D4 in human lung epithelial A549 cells. Ann Allergy Asthma Immunol. 2009 Oct;103(4):358-9. doi: 10.1016/S1081-1206(10)60540-6. No abstract available. PMID 19852204
- [Background] Schurman JV, Danda CE, Friesen CA, Hyman PE, Simon SD, Cocjin JT. Variations in psychological profile among children with recurrent abdominal pain. J Clin Psychol Med Settings. 2008 Sep;15(3):241-51. doi: 10.1007/s10880-008-9120-0. Epub 2008 Jul 25. PMID 19104969
- [Background] Tack J, Talley NJ, Camilleri M, Holtmann G, Hu P, Malagelada JR, Stanghellini V. Functional gastroduodenal disorders. Gastroenterology. 2006 Apr;130(5):1466-79. doi: 10.1053/j.gastro.2005.11.059. PMID 16678560
- [Background] Schurman JV, Singh M, Singh V, Neilan N, Friesen CA. Symptoms and subtypes in pediatric functional dyspepsia: relation to mucosal inflammation and psychological functioning. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):298-303. doi: 10.1097/MPG.0b013e3181d1363c. PMID 20479684
- [Background] Tusher VG, Tibshirani R, Chu G. Significance analysis of microarrays applied to the ionizing radiation response. Proc Natl Acad Sci U S A. 2001 Apr 24;98(9):5116-21. doi: 10.1073/pnas.091062498. Epub 2001 Apr 17. PMID 11309499
- [Background] Efron B, Tibshirani R, Storey JD, Tusher V. Empirical Bayes analysis of a microarray experiment. J Am Stat Assoc 2001;96:1151-1160.
- [Background] Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. J Royal Stat Soc Ser B 1995;57:289-300.
- [Background] Kazani S, Wechsler ME, Israel E. The role of pharmacogenomics in improving the management of asthma. J Allergy Clin Immunol. 2010 Feb;125(2):295-302; quiz 303-4. doi: 10.1016/j.jaci.2009.12.014. PMID 20159237